CLINICAL TRIAL: NCT02456038
Title: A Multicenter Study of the Safety and Efficacy of Asfotase Alfa (ALXN1215) (Human Recombinant Tissue Nonspecific Alkaline Phosphatase Fusion Protein) in Patients With Hypophosphatasia (HPP)
Brief Title: Safety and Efficacy of Asfotase Alfa in Patients With Hypophosphatasia (HPP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Osaka University Graduate School of Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HPPJEAP-01; UMIN000014816 (Other: UMIN CTR)
Record Dates: First submitted 2015-03-26; First posted 2015-05-28 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Hypophosphatasia
MeSH Terms: conditions — Hypophosphatasia | interventions — asfotase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Asfotase Alfa (ALXN1215) (Experimental): Asfotase Alfa (ALXN1215) is administered 6mg/kg in total per week, divided into 3 times.
  Interventions: Drug: Asfotase Alfa (ALXN1215)

INTERVENTIONS:
Drug: Asfotase Alfa (ALXN1215)
  Other Names: ALXN1215

SUMMARY:
The aim of this study is to assess safety and efficacy of Asfotase Alfa (ALXN1215) in patients with hypophosphatasia

ELIGIBILITY:
Inclusion Criteria:

Patients must meet one selection criteria of following "1", "2", and "3", and must meet the selection criteria of "4."

1. Patient who has been already treated with Asfotae Alfa (ALXN1215) out of this clinical trial
2. Patient who has been diagnosed as HPP
3. Documented diagnosis of HPP as indicated by:

<!-- -->

1. Total serum alkaline phosphatase below the lower limit of normal for age
2. Ultrasonographic features of prenatal, characterized by:

1) severe short extremities (femur length <-4SD in second and third trimesters) 2) extending into the metaphysis (femur metaphysis length or femur length >0.33) 3) craniotabes 4) Hypoplastic thorax (Thoracic or abdominal circumference <0.6) (3) Computed tomographic findings of prenatal, characterized by:

1. Generalized decreased ossification
2. Extreme shortening of tubular bones
3. Hypoplastic thorax (4) Radiographic evidence of HPP, characterized by:

1) Flared and frayed metaphyses 2) Severe, generalized osteopenia 3) Widened growth plates 4) Areas of radiolucency or sclerosis (5) Two or more of the following HPP-related findings:

1. History or presence of:

   - Nontraumatic post-natal fracture

   - Delayed fracture healing
2. Nephrocalcinosis or history of elevated serum calcium
3. Functional craniosynostosis
4. Respiratory compromise or rachitic chest deformity
5. Vitamin B6 dependent seizures
6. Failure to thrive
7. Premature tooth loss (6) Patient who have the mutation of tissue non-specific ALP gene 4. Parent or legal guardian(s) must provide written informed consent prior to any study procedures being performed and must be willing to comply with all study-required procedures

Exclusion Criteria:

1. Current evidence of treatable form of rickets
2. Serum calcium or phosphate levels below the normal range
3. Pregnant women and nursing mothers
4. Patient who cannot enforce suitable contraceptive measures during the clinical trial
5. Prior treatment with bisphosphonates
6. Treatment with an investigational drug within 1 month prior to the start of asfotase alfa treatment
7. Current enrollment in any other study involving an investigational new drug, device or treatment for HPP (e.g., bone marrow transplantation)
8. Clinically significant disease that precludes study participation, in the opinion of the Investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Adverse Events as an assessment of the Safety of repeated subcutaneous (SC) injections of asfotase alfa | Up to 50 months or until regulatory approval
  Safety of repeated subcutaneous (SC) injections of asfotase alfa for all treated patients

SECONDARY OUTCOMES:
Overall survival | Up to 50 months or until regulatory approval
  Overall survival is defined as the time from birth to time of death.
Effect of asfotase alfa treatment on skeletal manifestations of HPP as measured by radiographs using a qualitative Radiographic Global Impression of Change (RGI-C) scale | Up to 50 months or until regulatory approval
  Effect of asfotase alfa treatment on skeletal manifestations of HPP as measured by radiographs using a qualitative Radiographic Global Impression of Change (RGI-C) scale for all treated patients
Effect of asfotase alfa treatment on ventilator-free survival: (percentage of patients who are alive and ventilator-free after receiving asfotase alfa) | Up to 50 months or until regulatory approval
  For patients who are not mechanically ventilated at the time of enrollment, the percentage who are alive and ventilator-free after receiving asfotase alfa
Profile of asfotase alfa treatment on respiratory function | Up to 50 months or until regulatory approval
  Effect of asfotase alfa treatment on respiratory function as measured by ventilator status, time on respiratory support (including time on ventilator or supplemental oxygen), ventilator rate or oxygen volume, ventilator pressures, and fraction of inspired oxygen (FiO2) for all treated patients
Profile of asfotase alfa treatment on physical growth | Up to 50 months or until regulatory approval
  Effect of asfotase alfa treatment on physical growth as measured by body weight, length, arm span, head circumference, and chest circumference for all treated patients
Effect of asfotase alfa treatment on development | Up to 50 months or until regulatory approval
  Assessment of changes in gross motor development as measured by the developmental motor milestones for all treated patients

CONTACTS AND LOCATIONS:
Overall Officials: Keiichi Ozono, Principal Investigator — Osaka University Hospital
Locations (12):
- Japan (12):
  - Kurume University Hospital, Kurume, Fukuoka
  - National Hospital Organization Nagara Medical Center, Gifu, Gifu
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido-prefecture
  - Tohoku University Hospital, Sendai, Miyagi
  - Niigata University Medical & Dental Hospital, Niigata, Niigata
  - Osaka Medical Center and Research Institute for Maternal and Child Health, Izumi, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Saitama Children's Medical Center, Saitama, Saitama
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - Showa General Hospital, Kodaira, Tokyo